CLINICAL TRIAL: NCT04953429
Title: Correlation Between Workload and Sleep Quality of Shift Nurses in Top Three Hospitals in Beijing
Brief Title: Workload and Sleep Quality of Hospital Shift Nurses
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2020306
Record Dates: First submitted 2021-06-27; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-06

CONDITIONS: Workload; Sleep Quality
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Workload

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- nurses: nurses in a third-grade hospital in Beijing
  Interventions: Behavioral: workload

INTERVENTIONS:
Behavioral: workload — Mental needs, physical needs, time needs, self performance, effort, frustration, technical autonomy, decision-making autonomy and work needs of nursing work

SUMMARY:
A questionnaire survey was conducted to investigate the status of workload, sleep quality and the correlation between workload and sleep quality of shift nurses in Grade 3A hospitals in Beijing

DETAILED DESCRIPTION:
The shift nurses in the top three hospitals in Beijing were included. According to the sample size calculation method of correlation coefficient in analytical research, the correlation coefficient between workload and sleep quality was obtained by consulting literature ρ=- 29, confidence level α= 0.05, β= Then the sample size calculation software pass 11.0 was used to calculate n = 99. Considering 20% sample loss, the final sample size was n = 119. The same interviewee (head nurse / nurse) was informed of the purpose and significance of this study by using the same guiding language. The head nurses were informed one-on-one by the implementer of the project and filled in the questionnaire after informed consent; The nurse survey was conducted by the project implementer himself to the head nurse of the Department for training. The head nurse informed the nurses of the Department with unified guidelines, and after informed consent, the head nurse sent the electronic questionnaire QR code to its wechat work group for filling in. The implementer of the project will check the questionnaire in time after the respondents fill in the questionnaire, and give timely feedback if there is any doubt. This study investigated the work load and sleep quality of nurses in the top three hospitals in Beijing; The survey included general information, workload and sleep quality. General information included gender, age, working years, professional title, education level, marriage and childbearing status, etc. The workload status includes mental needs, physical needs, time needs, self performance, effort, frustration, technical autonomy, decision-making autonomy and work needs. The sleep quality status of nurses in different shifts (day shift, night shift and night shift) included sleep disorder, difficulty in maintaining sleep, early wake-up, fatigue / sleepiness in working days and idle time in working days, etc.

ELIGIBILITY:
Inclusion Criteria:

1. In service nurses who have obtained the nurse practice certificate of the people's Republic of China and have been registered;
2. At present, he has been involved in shift work for more than 3 months, and the shifts include day shift, night shift and night shift;
3. No obvious psychological or mental illness, such as depression; 4 volunteer to participate in this study.

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: nurses in a third-grade hospital in Beijing
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
sleep quality1 | 1 month
  Sleep disorders
sleep quality2 | 1 month
  difficulty in maintaining sleep
sleep quality3 | 1 month
  early awakening

CONTACTS AND LOCATIONS:
Overall Officials: Baohua Li, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No